CLINICAL TRIAL: NCT05983939
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Escalating Single and Multiple Doses of PIPE_791 and Food Effect in Normal Healthy Volunteers
Brief Title: Study Evaluating Safety and Tolerability of Escalating Single and Multiple Doses of PIPE-791 and Food Effect in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Contineum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PTI-791-101
Record Dates: First submitted 2023-07-19; First posted 2023-08-09 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; PIPE-791; Health volunteers
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All roles are masked with the exception of the pharmacist/dose preparer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PIPE-791 (Experimental)
  Interventions: Drug: PIPE-791
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PIPE-791 — Single and multiple ascending oral doses of PIPE-791 tablets.
  Arms: PIPE-791
Drug: Placebo — Single and multiple ascending oral doses of matching placebo tablets.
  Arms: Placebo

SUMMARY:
This study will be conducted in three parts: Part 1 will be a Single Ascending Dose (SAD), Part 2 will be a Multiple Ascending Dose (MAD), and Part 3 will be a selected SAD cohort in a fed state. Safety will be assessed by periodic measurement of vital signs, physical examinations, electrocardiograms, blood laboratory analyses and occurrence of adverse events (AE).

DETAILED DESCRIPTION:
This is a randomized, double-blind study of PIPE-791 or placebo given as single and multiple escalating doses in normal healthy subjects. The study will be conducted in three parts: Part 1 will be a Single Ascending Dose (SAD) study enrolling approximately 48 subjects for a total duration of 6 weeks. Part 2 will be a Multiple Ascending Dose (MAD) study enrolling approximately 32 subjects for a total duration of 7 weeks, and part 3 will be a selected SAD cohort in a fed state to evaluate the effect of food on the bioavailability of PIPE-791, enrolling approximately 8 subjects for a duration of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age (inclusive) at the time of signing informed consent.
* Male or female subjects with reproductive potential agree to comply with protocol-approved double barrier contraceptive method 30 days prior to the first dose and up to 90 days post last dose.
* Medically healthy with no clinically significant or relevant abnormalities in medical history, physical exam, vital signs, electrocardiogram (ECG), or laboratory evaluations (hematology, chemistry, and urinalysis) as assessed by the Investigatory.

Exclusion Criteria:

* Has a current or recurrent disease that could affect the investigational medicinal product or affect clinical or laboratory assessments.
* Experienced a significant systemic illness, as judged by the Investigator, within 30 days of the first dose.
* Has a history of a significant medical, including hepatic and/or renal disease as outlined in the protocol, or psychiatric disorder that may require treatment or make the participant unlikely to fully complete the study or increase risk to the participant.
* History of alcohol or other substance abuse within the 12 months prior to the dosing at the discretion of the Investigator.
* Routine alcohol consumption meeting or exceeding protocol limits.
* History of prior malignancy (except adequately treated non-melanoma skin cancer, carcinoma in-situ of the uterine cervix, ductal carcinoma in situ (DCIS), or localized prostate cancer).
* Donated or lost more than 400 mL of blood within 56 days or plasma within 14 days prior to Screening.
* Received an investigational agent within the last 30 days, prior to screening, or five half-lives of the prior investigational agent.
* Use of any prescription medication, over-the-counter medication, vitamin or supplement, herbal or homeopathic preparation within 7 days or 5 half-lives prior to study drug administration, as determined by the Investigator. Hormone replacement therapy and hormonal contraception is permissible throughout the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Safety: Treatment-Emergent Adverse Events (TEAE) | Baseline to 14 days post dosing for SAD cohorts and 14 days post dosing for MAD cohorts
  Number of participants with TEAEs

SECONDARY OUTCOMES:
Safety: Cardiac repolarization using Fridericia-corrected QT interval (QTcF) | Baseline to 14 days post dosing for SAD cohorts and 14 days post dosing for MAD cohorts
  Change in mean QTcF
Pharmacokinetics (PK): Blood concentration levels of PIPE-791 | Baseline to 14 days post dosing for SAD cohorts and 14 days post dosing for MAD cohorts
Pharmacokinetics: Urine concentration levels of PIPE-791 | Baseline on day 1 through day 2 for SAD cohorts and from baseline on day 1 through day 7 for MAD cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Huhn, MD, Study Director — Pipeline Therapeutics
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No